CLINICAL TRIAL: NCT02379754
Title: Gentamicin Treatment Prior to Vestibular Schwannoma Surgery in Patients With Definite Remaining Vestibular Function
Brief Title: Gentamicin Treatment Prior to Schwannoma Surgery - Residual Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VS-FT-01
Record Dates: First submitted 2015-01-25; First posted 2015-03-05 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Vestibular Schwannoma
Keywords: vestibular schwannoma; acoustic neuroma; cerebellopontine angle tumour; gentamicin; rehabilitation; postural balance
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gentamicin treated (Experimental): Installation of gentamicin in the middle ear 6 weeks prior to surgery + rehabilitation exercises before and after both treatment and surgery.
  Rehabilitation exercises are not considered to be an intervention since their benign impact on vestibular/postural compensation is well documented, and exclusion from exercises would not be approved by the ethical board.
  Interventions: Drug: Gentamicins
- Non-gentamicin (No Intervention): Rehabilitation exercises before and after surgery. Rehabilitation exercises are not considered to be an intervention since their benign impact on vestibular/postural compensation is well documented, and exclusion from exercises would not be approved by the ethical board.

INTERVENTIONS:
Drug: Gentamicins — Intratympanic installation of gentamicin 2-4 times depending on the efficacy of vestibular deafferentation
  Other Names: Prehabituation, PREHAB; Intratympanic installation of gentamicin
  Arms: Gentamicin treated

SUMMARY:
The purpose of the study is to determine whether vestibular and postural compensation following schwannoma surgery is improved by ablating remaining vestibular function prior to surgery, through gentamicin injections in the middle ear.

DETAILED DESCRIPTION:
The residual function of the vestibular system before surgery differs considerably between patients, due to extent and influence of tumor growth, resulting in varying spectra of post-surgery illness as well as vestibular symptoms. An acute unilateral vestibular deafferentation (uVD) (if significant vestibular function remains prior to surgery) invariably results in severe nausea and vertigo. The nausea/vertigo induced by surgery and sudden uVD both can impede vestibular compensation processes and in extension, also the need for rehabilitation. The vestibular PREHAB protocol was developed in order to address this problem and to ensure an enhanced and sufficient rehabilitation. The protocol encompass treating patients that have measurable vestibular function before surgery with intratympanic gentamicin injections, thus producing gradually a uVD over a period of 3-4 weeks, whilst performing daily vestibular exercises before and after the gentamicin treatment. Through this procedure the sensory trauma is separated from the surgical trauma, making it possible for vestibular compensation to ensue as the vestibular function gradually decline from gentamicin toxicity, unencumbered by any depression of central nervous function that might result from schwannoma surgery or the acute stages of an uVD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with vestibular schwannoma and surgical treatment is advised
* remaining vestibular function

Exclusion Criteria:

* impaired decision making
* no remaining vestibular function
* signs of central nervous dysfunction
* neurofibromatosis
* Patients are advised not to participate in the gentamicin arm but encouraged to participate in the 'non-gentamicin' arm:
* when hearing is better than 30decibel (dB) i pure tone average (500, 1000, 2000, 3000/4000 Hz) and speech discrimination better than 70% -when the neurosurgeon aim at hearing preservation surgery and do not want to risk gentamicin- associated hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2019-06 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Differences and changes of postural control following surgery, compared to before surgery | At first vestibular assessment at the time for inclusion and 6 months after surgery
  Postural control assessed with posturography during a sensory conflict

SECONDARY OUTCOMES:
Differences of duration of hospital stay | After surgery for the duration of the hospital stay up to two weeks
  Hospital stay required before patients can be discharged
Differences of subjective well being after surgery | Immediate time after surgery (2 weeks)
  Daily subjective assessment of perceived vertigo/dizziness after surgery and gentamicin treatment
Change of subjective well being after gentamicin treatment | Immediate time after gentamicin installation (2 weeks)
  Daily subjective assessment of perceived vertigo/dizziness after gentamicin treatment
Change of hearing levels | At first vestibular assessment and 2 weeks after gentamicin installation
  Measuring hearing levels (pure tone hearing and speech discrimination) before and after gentamicin treatment to determine possible detrimental effect on hearing
Differences in the level of stress after surgery | Daily after surgery for the duration of the hospital stay up to 2 weeks
  Daily Measures of cortisol in the saliva after surgery during the time patients are admitted to the hospital
Differences of perceived dizziness after surgery | 6 months after surgery
  Measure of level of impact of dizziness in daily life, measured with Dizziness Handicap Inventory (DHI)
Differences of level of anxiety and depression | 6 months after surgery
  Measure of level of anxiety and depression after surgery, enquiry with Hospital Anxiety and Depression Scale (HADS)
Change of level of perceived dizziness after gentamicin | At first vestibular assessment and 6 weeks after gentamicin installation
  Measure of level of impact of dizziness in daily life, measured with Dizziness Handicap Inventory (DHI)
Differences of changes in levels of perceived dizziness after surgery as compared to before surgery | At first vestibular assessment and 6 months after surgery
  Measure of level of impact of dizziness in daily life, measured with Dizziness Handicap Inventory (DHI)
Occurrence of spontaneous nystagmus after surgery | Day 1 after surgery and for duration of either spontaneous nystagmus or hospital stay (up to 2 weeks)
  To measure spontaneous nystagmus after surgery and its direction as a sign of vestibular deafferentation or central nervous damage
Differences in vestibular compensation after surgery | 6 months after surgery
  Vestibular function tests, v-HIT, calorics and otolith tests to determine compensation after surgery
Change of vestibular function after gentamicin treatment | 6weeks after gentamicin treatment
  Vestibular function tests, v-HIT, calorics and otolith tests to determine compensation and function after gentamicin treatment

OTHER OUTCOMES:
Differences of needed sick-leave from work and leisure activities | 6 months after surgery
  Time to return to normal daily activities after surgery, both job-related and leisure activities

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Tjernström, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Dept. OtoRhinoLaryngology Head and Neck Surgery, Skane University Hospital, Lund, Sweden

REFERENCES:
- [Background] Magnusson M, Padoan S. Delayed onset of ototoxic effects of gentamicin in treatment of Meniere's disease. Rationale for extremely low dose therapy. Acta Otolaryngol. 1991;111(4):671-6. doi: 10.3109/00016489109138398. PMID 1950529
- [Result] Tjernstrom F, Fransson PA, Kahlon B, Karlberg M, Lindberg S, Siesjo P, Magnusson M. Vestibular PREHAB and gentamicin before schwannoma surgery may improve long-term postural function. J Neurol Neurosurg Psychiatry. 2009 Nov;80(11):1254-60. doi: 10.1136/jnnp.2008.170878. Epub 2009 Jul 1. PMID 19574236
- [Result] Magnusson M, Kahlon B, Karlberg M, Lindberg S, Siesjo P, Tjernstrom F. Vestibular "PREHAB". Ann N Y Acad Sci. 2009 May;1164:257-62. doi: 10.1111/j.1749-6632.2009.03778.x. PMID 19645909
- [Result] Magnusson M, Karlberg M, Tjernstrom F. 'PREHAB': Vestibular prehabilitation to ameliorate the effect of a sudden vestibular loss. NeuroRehabilitation. 2011;29(2):153-6. doi: 10.3233/NRE-2011-0689. PMID 22027076
- [Result] Magnusson M, Kahlon B, Karlberg M, Lindberg S, Siesjo P. Preoperative vestibular ablation with gentamicin and vestibular 'prehab' enhance postoperative recovery after surgery for pontine angle tumours--first report. Acta Otolaryngol. 2007 Dec;127(12):1236-40. doi: 10.1080/00016480701663433. PMID 17917842
- [Result] Postema RJ, Kingma CM, Wit HP, Albers FW, Van Der Laan BF. Intratympanic gentamicin therapy for control of vertigo in unilateral Menire's disease: a prospective, double-blind, randomized, placebo-controlled trial. Acta Otolaryngol. 2008 Aug;128(8):876-80. doi: 10.1080/00016480701762458. PMID 18607963